CLINICAL TRIAL: NCT06296082
Title: Comparative Study of the Mechanism of Action of Dry Needling and Botulinum Toxin Type A as a Treatment for Lower Limb Post-stroke Spasticity: a Proof of Concept Controlled Trial
Brief Title: Comparative Study of the Effects of Dry Needling and Botulinum Toxin Type A as a Treatment for Lower Limb Post-stroke Spasticity
Acronym: STROKEPOC
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Instituto de Investigación Sanitaria Aragón (Other); McGill University (Other); Instituto de Salud Carlos III (Other Government); Fonds de la Recherche en Santé du Québec (Other Government); Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Dr. Pablo Herrero Gallego, Prof. Dr., Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 49317
Record Dates: First submitted 2024-02-13; First posted 2024-03-06 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Stroke
Keywords: Stroke [Mesh]; Dry Needling; Muscle Spasticity [Mesh]; Botulinum Toxins [Mesh]; Tonic Stretch Reflex Threshold; Ultrasound imaging; Gait analysis; Quality of Life [Mesh]
MeSH Terms: conditions — Stroke | interventions — Botulinum Toxins, Type A; Dry Needling

STUDY DESIGN:
Intervention Model Description: A prospective randomized, controlled, multiple-baseline, and assessor blinded multicenter equivalence trial with two parallel groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessments will be conducted by blinded assessors for treatment allocation. Participants and staff cannot be blinded due to the nature of the intervention, but are instructed not to disclose their treatment allocation. Data will be anonymized and an independent researcher will enter coded data into secure databases. Data will be analyzed by a blinded statistician. Code breaks will only be allowed in crucial cases for patient management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Botulinum Toxin type A (Active Comparator): The BTX-A group will receive onabotulinumtoxinA (Botox®, Allergan) with mandatory muscles getting 300 units and optional muscles getting up to 100 additional units (maximum dose of 400 units) (14) delivered with a 27-gauge (0.45 mm) beveled needle. Target muscles will be identified by ultrasound imaging or muscle stimulation. Local anesthesia will not be used. Patient positioning will be standardized.
  Interventions: Drug: Botulinum toxin type A
- Dry Needling (Active Comparator): For Dry Needling group solid, filiform non-beveled 0.30 mm caliber needles will be used. Target muscles will be identified by ultrasound imaging or muscle stimulation. Local anesthesia will not be used. Patient positioning will be standardized.
  Interventions: Other: Dry Needling

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum toxin type A injections are a treatment technique to treat the spastic muscles in patients with stroke that targets on the neuromuscular endplate zone provoking a chimical disruption of dysfunctional endplates.
  Arms: Botulinum Toxin type A
Other: Dry Needling — Dry Needling is a treatment technique to treat the spastic muscles in patients with stroke that targets on the neuromuscular endplate zone provoking a mechanical disruption of dysfunctional endplates.
  Arms: Dry Needling

SUMMARY:
This is a randomized parallel group clinical trial which will be conducted in three countries (Spain, Canada and Belgium) comparing Botulinum Toxin type A (BTX-A) and Dry Needling (DN) effectiveness for post-stroke spasticity in participants who had a first stroke in the previous 12 months and have plantar flexor spasticity. Participants will be randomly allocated to receive either one session of BTX-A or 12 weekly sessions of DN. Blinded evaluators will assess the effects before, during, and after treatment, and at a 4-week follow-up.

DETAILED DESCRIPTION:
The primary hypothesis is that the effects of DN on post-stroke spasticity in the lower limbs at the spinal level is comparable to BTX-A in reducing spasticity by decreasing stretch reflex excitability.

Sample size: Spain, Canada and Belgium will recruit 90 participants (30 per country)

The platform used for randomization and electronic data collection will be Research Electronic Data Capture (REDcap): https://www.project-redcap.org/. A shared license will be used among the countries involved in the study.

Data dictionary:

* DN: Dry Needling
* BTX-A: Botulinum toxin type A
* TSRT: Tonic Stretch Reflex Threshold
* MAS: Modified Ashworth Scale
* 10MWT: 10 Metre Walk Test
* TUG: Timed Up & Go
* PPI: Public and Patient Involvement
* SOP: Standard Operating Procedure

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-75 years.
2. post-stroke spasticity in ankle plantar flexors (Modified Ashworth Scale (MAS) scores of 1-2).
3. first stroke.
4. 0-12 months evolution.
5. no previous BTX-A or DN treatment for spasticity.
6. ankle passive range of motion ≥ 20° (approximately) with knee flexion ~30°.
7. independent ambulation with or without aids.

Exclusion Criteria:

1. medical conditions interfering with data interpretation.
2. contraindications for BTX-A or DN treatment.
3. changes in anti-spasticity medication dosage (if appropriate), either during the trial or within the 3 months prior to participation.
4. pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tonic Stretch Reflex Threshold (TSRT) | Week 1 to 15 and 19.
  TSRT is a novel measures of stretch reflex excitability that provide an indirect indicator of the excitability of α-motoneurons at the level of the spinal cord.

SECONDARY OUTCOMES:
Muscle thickness | Week 1 to 15 and 19.
  It is the estimation of the thickness of the muscle fiber, which is obtained by tracing a line that covers the length of the muscle between the deep and superficial aponeuroses.
Pennation angle | Week 1 to 15 and 19.
  It is the angle between the deep fascia and the line of the fascicle length.
Concurrence matrices | Week 1 to 15 and 19.
  Measures that describe the spatial distribution of gray levels in the texture of an ultrasound image. These matrices, also known as co-occurrence matrices, are used to analyze textural features and patterns in ultrasound images.
Resistance to passive stretching | Week 1 to 15 and 19.
  It will be measured using the Modified Ashworth Scale (MAS). The scale ranges from a minimum value of 0 to a maximum of 4, with 0 indicating no spasticity (no resistance to passive stretching) and 4 representing the most severe spasticity (resistance to passive stretching), characterized by complete rigidity.
Gait analysis | Week 1,2,9,15 and 19
  It will be done with motion capture systems using wearable and inertial sensors. Canada and Belgium: Xsens system (MVN Awinda, Movella, Hendersen, USA); Spain: Move Human Sensors MoCap System.
Functional mobility | Week 1,2,9,15 and 19
  Measured by Time Up and Go (TUG).
Functional mobility | Week 1,2,9,15 and 19
  Measured by 10 Meter Walk Test (10MWT)
Muscle Strength | Week 1 to 15 and 19.
  Muscle strength will be measured by hand-held dynamometry (MicroFET 2)
Quality of life analysis | Week 1, 15 and 19.
  It will be assessed with the EuroQOL-5D (Euro Quality of Life-5 Dimensions-5 Levels). Responses from the questionnaire will be converted to health-state utility values, where higher values represent improved quality of life. Index scores range from -0.59 to 1, where 1 is the best possible health state.
Cost-effectiveness | Week 19.
  Costs related to treatment will be assessed by computing the ICER (Incremental cost-effectiveness ratio) in €/QALY (Quality-Adjusted Life Year)
Safety: Frequency and severity of Dry Needling (DN) and Botulinum Toxin type A (BTX-A) adverse events | Week 3 to 14 and 19.
  Description of the adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Herrero Gallego, PhD, Principal Investigator — Universidad de Zaragoza
Locations (3):
- Universiteit Antwerpen, Antwerp, Flanders, Belgium
- Jewish Rehabilitation Hospital, Montreal, Quebec, Canada
- Hospital Clínico Universitario Lozano Blesa, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared with other researchers in accordance with data sharing protocols and participant consent, ensuring confidentiality and ethical considerations are maintained.
Supporting Information: Study Protocol
Time Frame: Data will be available for 15 years.
Access Criteria: In relation to other academic institutions and in the possession of a Good Clinical Practice Certificate

REFERENCES:
- See also: Web site of the project. — https://www.itonus.eu/